CLINICAL TRIAL: NCT05910398
Title: Continuous or Intermittent Extension of Adjuvant Pyrotinib for Invasive Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Breast Cancer: a Prospective, Randomised, Controlled, Multicentre Clinical Trial
Brief Title: Continuous or Intermittent Extension of Adjuvant Pyrotinib for Invasive HER2-positive Breast Cancer
Acronym: CORINNE-PI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LY2023-063-A
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Invasive
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continuous pyrotinib (Active Comparator): pyrotinib 400 mg, orally once daily for one year
  Interventions: Drug: pyrotinib
- intermittent pyrotinib (Experimental): pyrotinib 400 mg, 14 days on and 7 days off, every 21 days for 17 cycles
  Interventions: Drug: pyrotinib

INTERVENTIONS:
Drug: pyrotinib — an irreversible anti-HER2 tyrosine kinase inhibitor

SUMMARY:
This is a prospective, randomised, controlled, multicentre study to compare the efficacy and safety between continuous or intermittent extension of adjuvant pyrotinib in invasive human epidermal growth factor receptor 2 (HER2)-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18;
* Histologically confirmed invasive HER2 positive breast cancer;
* Duration from random time to the last use of trastuzumab or T-DM1 ≤3 years;
* Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1;
* Adequate organ functions.

Exclusion Criteria:

* Metastatic disease (Stage IV);
* Gross residual disease remaining after mastectomy or positive margins after breast-conserving surgery;
* Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption;
* Treated or treating with anti-HER2 tyrosine kinase inhibitor;
* Less than 4 weeks from the last clinical trial;
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation;
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test; Female patients of childbearing age that are reluctant to take effective contraceptive measures throughout the trial period;
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (iDFS) | From randomization until time of event up to 2 years.
  Invasive disease-free survival time is defined as the time from date of randomization until the first invasive disease recurrence of the following events: invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, distant recurrence and death from any cause.

SECONDARY OUTCOMES:
Disease-free Survival (DFS) | From randomization until time of event up to 2 years
  Disease-free survival time is defined as the time from date of randomization until the first disease recurrence of the following events: invasive ipsilateral breast tumor recurrence, invasive contralateral breast cancer, local/regional invasive recurrence, non-breast primary invasive cancer, ductal carcinoma in situ (DCIS),or distant recurrence and death from any cause
Overall Survival (OS) | From randomization until time of event up to 2 years
  Overall survival is defined as the time from randomization to death from any cause.
Adverse events | From the date of starting pyrotinib to the end of the treatment (up to approximately 1 year)
  Adverse events will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No